CLINICAL TRIAL: NCT03703492
Title: Positron Emission Tomography/Magnetic Resonance Imaging of Estrogen Receptor Expression n Non-Invasive Breast Cancer
Brief Title: Hybrid Molecular Imaging of ER in Breast Cancer Patients With DCIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UW18063; KL2TR000428 (NIH); NCI-2018-02281 (Registry Identifier: NCI Trial ID); 2018-0814 (Other: Institutional Review Board); A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); P30CA014520 (NIH); Protocol Version 5/11/2022 (Other: UW Madison)
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ - Category
MeSH Terms: conditions — Breast Neoplasms | interventions — 16-fluoroestradiol; gadobenic acid

STUDY DESIGN:
Intervention Model Description: This is a prospective, one-arm, observational study which will enroll participants with biopsy-proven DCIS scheduled for diagnostic breast MRI for preoperative staging/extent of disease evaluation as part of standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Research Arm (Experimental): Directed breast PET/MRI with 18F-FES; 18F-FES uptake of the known malignancy to be measured on the PET/MRI examination
  Interventions: Drug: (18F)FES; Drug: Gadobenate dimeglumine

INTERVENTIONS:
Drug: (18F)FES — 18F-FES is an investigational new drug which will be used for this study. For complete information, please refer to the Investigator's Brochure: "[18F]Fluoroestradiol: An investigational positron emission tomography (PET) radiopharmaceutical for injection, intended for use as an in vivo diagnostic for imaging estrogen receptors in tumors
  Other Names: 11.2 16α-[18F]-fluoro-17β-estradiol; FES
Drug: Gadobenate dimeglumine — Gadolinium-based intravenous contrast agent used for the MRI portion of this study
  Other Names: MultiHance

SUMMARY:
This prospective, one-arm study which will enroll participants with biopsy-proven DCIS scheduled for diagnostic breast MRI for preoperative staging/extent of disease evaluation as part of standard of care. Eligible participants will be consented for participation in the research study which includes a directed breast PET/MRI with 18F-FES. 18F-FES uptake of the known malignancy will be measured on the PET/MRI examination using standardized uptake values (SUV) and tumor-to-normal tissue ratios.

DETAILED DESCRIPTION:
Integrated whole-body magnetic resonance imaging (MRI)-positron emission tomography (PET) scanners have recently been introduced for clinical use. This technology combines the anatomic and perfusion data obtained with Dynamic Contrast Enhanced (DCE) MRI with functional imaging data obtained from PET. For breast imaging, the combination of MRI and PET has important potential to improve diagnostic accuracy and provide molecular characterization of breast cancer. The overall purpose of this research is to determine the technical feasibility of simultaneous breast DCE MRI with 18F-FES PET for measuring estrogen receptor (ER) in patients with ductal carcinoma in situ (DCIS) and identifying patients with low-risk of disease recurrence. The hypothesis is that quantitative 18F-FES uptake parameters from PET/MRI will correlate well with the ER immunohistochemistry score and with low-risk recurrence scores.

Primary Objective 1) To compare quantitative 18F-FES uptake of biopsy-proven DCIS measured using PET/MRI with ER protein levels determined by immunohistochemistry.

Secondary Objectives

1. To determine the optimal cut-point 18F-FES uptake value for distinguishing between ER+ and ER-negative DCIS
2. To determine the test-retest reproducibility of quantitative assessment of tumor 18F-FES uptake
3. To determine the optimal cut-point 18F-FES uptake value for distinguishing between low-risk DCIS and intermediate/high-risk DCIS
4. To estimate the association of quantitative 18F-FES uptake (continuous SUVmax) with research-based Oncotype DX DCIS scores (0-100)
5. To measure the upgrade rate to invasive cancer at surgical excision
6. To correlate tumor 18F-FES uptake with serum estradiol and sex hormone binding globulin levels.

Exploratory Objective

1) To correlate tumor cell density with 18F-FES uptake on PET/MRI

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of biopsy-proven DCIS without invasion or microinvasion measuring at least 1.0 cm in diameter by any imaging modality
* Undergoing diagnostic breast MRI ordered by the referring clinician for staging and extent of disease

Exclusion Criteria:

* Inability or unwillingness to provide informed consent to the study
* Surgery, radiation, neoadjuvant chemo/endocrine therapy for the current malignancy prior to study enrollment
* Participants currently taking or have taken an ER-blocking medication (e.g. tamoxifen, raloxifene) within 6 weeks prior to study enrollment
* Pregnant or lactating women
* Participant with intolerance or contraindications for MRI or gadolinium-based contrast agents
* Participant girth exceeds the bore of the MRI/PET scanner
* Participants with a history of allergic reaction attributable to compounds of similar chemical or biologic composition to 18F-FES
* Participants in liver failure as judged by the patient's physician, due to the hepatobiliary clearance of 18F-FES
* Participants requiring intravenous (IV) conscious sedation for imaging are not eligible; participants requiring mild, oral anxiolytics for the clinical MRI will be allowed to participate as long as the following criteria are met:

  * The participant has their own prescription for the medication
  * The informed consent process is conducted prior to the self-administration of this medication
  * They come to the research visit with a driver or an alternative plan for transportation (e.g. Uber, taxi, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Fowler, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at UW Health from January 2019 to December 2023.
Period: Overall Study
Arm/Group | Research Arm
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Research Arm
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  40 to 49 years old | 5
  50 to 59 years old | 5
  60 to 69 years old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: 18F-FES Uptake in DCIS
Description: 18F-FES uptake of biopsy-proven ductal carcinoma in situ (DCIS) measured using PET/MRI will be reported in Standardized Uptake Values (SUV).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Research Arm
Number analyzed (Participants) | 12
SUV | 1.43 (0.83)

2. Secondary Outcome: Prognostic Risk Categories Determined Using Van Nuys Prognostic Index, the MSKCC Nomogram
Description: ROC curve analysis will be performed to determine the optimal cut-point for 18F-FES SUVmax to distinguish low-risk DCIS and intermediate/high-risk DCIS. Risk categories will be determined using the Van Nuys Prognostic Index, the Memorial Sloan-Kettering Cancer Center Nomogram, and the research-based Oncotype DX DCIS score. Sensitivity and specificity will be determined with two-sided 95% confidence intervals. The area under the curve (AUCs) for the ROCs and their respective two-sided 95% confidence intervals will be calculated using logistic regression.
  The optimal cut-off point will be determined by considering the 18F-FES uptake value with the maximum sensitivity and specificity.
  This analysis will be done separately for each risk assessment model.
Time Frame: 2 months
Population: Data for low-risk DCIS is insufficient to perform ROC curve analysis.
Measure: Number (95% Confidence Interval); unit: AUC
Arm/Group | Research Arm
Number analyzed (Participants) | 12
AUC | NA [NA to NA] — Lack of events

3. Secondary Outcome: Research-based Oncotype DX DCIS Scores
Description: To estimate the association of quantitative 18F-FES uptake (continuous SUVmax) with research-based Oncotype DX DCIS scores (0-100), scatter plots of continuous quantitative 18F-FES uptake (SUVmax) on the y-axis and research-based Oncotype DX DCIS scores (unitless) on the x-axis will be created to explore the distribution of the measurements. Pearson's or Spearman's rank correlation will be used to evaluate the association between quantitative 18F-FES uptake and research-based Oncotype DX DCIS score. The correlation coefficient (rho) and 95% confidence interval will be reported.
Time Frame: 12 months
Population: There was not enough amount of RNA starting material from the samples to perform the assay. No data was collected for this outcome since the research-based assay could not be performed due to insufficient RNA isolation.
Arm/Group | Research Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Invasive Cancer at Surgical Excision
Description: This percentage will be calculated by dividing the number of patients with invasive breast cancer diagnosed at the time of surgical excision by the number of patients with percutaneous biopsy-proven DCIS in the study.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Research Arm
Number analyzed (Participants) | 12
Participants | 2

5. Secondary Outcome: Serum Estradiol Levels
Description: Mean serum estradiol levels will be reported to summarize the outcome measure.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Research Arm
Number analyzed (Participants) | 12
picograms per milliliter (pg/mL) | 31.3 (46.0)

6. Secondary Outcome: Serum Sex Hormone Binding Globulin Levels
Description: A correlation analysis of sex hormone binding globulin levels will be performed using Pearson's or Spearman's rank correlation. Scatter plots, correlation coefficients (rho) and 95% confidence intervals will be reported.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Research Arm
Number analyzed (Participants) | 12
nanomoles per liter (nmol/L) | 64.4 (43.0)

ADVERSE EVENTS:
Time Frame: up to 24 hours
Arm/Group | Research Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Research Arm (N=12)
IV site pain during injection (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03703492/Prot_SAP_000.pdf